CLINICAL TRIAL: NCT06711094
Title: Single-arm,Exploratory Clinical Study of Albumin-bound Paclitaxel Combination With Dalpiciclib and AI in the Treatment of ER-Low (1%-10%), HER2-negative Advanced Breast Cancer
Brief Title: Albumin-bound Paclitaxel、Dalpiciclib and AI in ER-Low (1%-10%) HER2-ABC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Fan Wu, Clinical Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fujian Cancer Hospital
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: HR+/HER2- Advanced Breast Cancer
MeSH Terms: interventions — dalpiciclib

STUDY DESIGN:
Intervention Model Description: prospective, single-arm, single-center, open, exploratory clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): albumin-bound paclitaxel、Dalpiciclib and AI
  Interventions: Drug: Dalpiciclib

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib: 125mg orally, with a treatment cycle every 28 days, with continuous administration for the first 3 weeks (days 1 to 21) and rest (no medication) for the second 1 week (days 22 to 28). It is recommended to take Dalpiciclib at about the same time every day.
  Albumin-bound paclitaxel for injection: 125mg/m2, intravenous infusion for 30 minutes, D1, D8, every 28 days for a treatment cycle, at least ≥6 treatment courses.
  Endocrine therapy: Endocrine therapy drugs are selected by the investigator

SUMMARY:
This is a prospective, single-arm, single-center, open, exploratory clinical study.. Screening for histopathologically confirmed recurrent or metastatic ER-Low positive (1%-10%) and HER2-negative breast cancer patients who meet the inclusion criteria and have not previously received any systemic anticancer therapy for advanced disease, He was treated with albumin-bound paclitaxel in combination with Dalpiciclib and AI.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center, open, exploratory clinical study. Simon two-stage sample size calculation was used in this study, and the primary endpoint was objective response rate (ORR). P0=37.3% (POLAMA-4 experimental group data), P1=53.2%, unilateral α=0.05, 1-β=80% were set. PASS15 software was used to calculate 21 cases in the first stage, with a total sample size of 52 cases. If 8 patients in Phase I achieve an objective response, proceed to Phase II. Screening for histopathologically confirmed recurrent or metastatic ER-Low positive (1%-10%) and HER2-negative (IHC 0/1+ or IHC 2+ but ISH-) breast cancer patients who meet the inclusion criteria and have not previously received any systemic anticancer therapy for advanced disease, He was treated with albumin-bound paclitaxel in combination with Dalpiciclib and AI.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal or premenopausal/perimenopausal women ≥18 years old and ≤75 years old, meeting one of the following criteria: a) prior bilateral oophorectomy, or ≥60 years old; Or b) age <60, natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH at postmenopausal levels; Or c) premenopausal or perimenopausal women may also be enrolled, but must be willing to receive LHRH agonist therapy during the study period.
2. Female breast cancer patients diagnosed by pathology as ER-Low positive (1%-10%) and HER2-negative have evidence of focal recurrence or metastasis, and are not suitable for surgical resection or radiotherapy for the purpose of cure. a) Low ER expression was defined as: the proportion of tumor cells with positive staining accounted for ≥ 1% and ≤10% of all tumor cells (confirmed by investigators in the study center); b) HER2 negative is defined as a standard immunohistochemical (IHC) test of 0/1+; Or the IHC test is 2+ and the ISH test is negative (reviewed and confirmed by the investigator at the study center).
3. Have not previously received any systemic anticancer therapy for recurrent or metastatic disease.
4. The physical status score of the Eastern Cancer Collaboration Group (ECOG) was 0-1.
5. Measurable lesions or bone metastases only (including osteolytic lesions or mixed osteolytic/osteoblastic lesions) that meet RECIST 1.1 criteria.
6. Adequate organ and bone marrow function.
7. Women of reproductive age must have a negative serum pregnancy test within 7 days prior to enrollment and be willing to use a medically approved highly effective contraceptive during the study period and within 3 months after the last study drug administration.
8. Remission of all acute toxic reactions from previous antitumor therapy to grade 0-1 (according to NCICTCAE version 5.0) or to the level specified in the inclusion/exclusion criteria. The exception is other toxicities, such as hair loss, that researchers believe do not pose a safety risk to patients.

Exclusion Criteria:

1. Previous pathological examination diagnosed HER2-positive breast cancer.
2. Inflammatory breast cancer.
3. Disease progression or recurrence during prior adjuvant therapy or within 12 months after completion of adjuvant therapy.
4. Patients judged unsuitable for chemotherapy by the investigators. This includes symptomatic, advanced patients who have spread to the viscera and are at risk of developing life-threatening complications in the short term (including patients with uncontrolled exudation [thoracic, pericardial, abdominal], pulmonary lymphangitis, and more than 50% liver involvement).
5. Patients with symptomatic active brain metastases or meningeal metastases were confirmed by cranial CT or MRI.
6. Previous treatment with any CDK4/6 inhibitors.
7. Major surgery, chemotherapy, radiation therapy, any investigational drug, or other anti-cancer treatment within 2 weeks prior to study entry.
8. Any other malignant tumor diagnosed within 3 years prior to study entry, except for non-melanoma skin cancer, basal cell or squamous cell skin cancer, or cervical carcinoma in situ after radical treatment.
9. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥1000 IU/ml), hepatitis C (HCV antibody positive and HCV-RNA above the lower detection limit of analytical methods), or co-infection with hepatitis B and hepatitis C.
10. Within 6 months prior to entering the study, the following situations occurred: Myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac insufficiency, persistent arrhythmias ≥ grade 2 (according to NCI CTCAE 5.0), atrial fibrillation of any grade, coronary/peripheral artery bypass surgery, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism).
11. Severe infection within 4 weeks prior to the first dose (e.g. intravenous antibiotic, antifungal, or antiviral medication required according to clinical practice), or unexplained fever >38.5°C during screening/prior to the first dose.
12. Inability to swallow, intestinal obstruction, or other factors affecting the administration and absorption of medications.
13. Known allergy to albumin-bound paclitaxel, letrozole, anastrozole, Metrotan, LHRH agonists (goserrelin, leprerelin), Darcilil, or any excipients.
14. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
15. Known history of psychotropic substance abuse or drug use.
16. The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participation in the study or interfere with the study results, as well as patients deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 2 year
  To assess and compare objective response rate (ORR) using RECIST 1.1

SECONDARY OUTCOMES:
PFS | through study completion, an average of 2 year
  To assess and compare efficacy by progression-free survival (PFS) using Response Evaluation Criteria In Solid Tumors 1.1 [RECIST 1.1]

IPD SHARING:
Plan to Share IPD: No